CLINICAL TRIAL: NCT01137565
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AMG 853 in Adolescent (≥ 12 to <18 Years) and Adult Subjects With Intermittent or Mild to Moderate Persistent Asthma
Brief Title: Safety, Tolerability, and Pharcodynamics of AMG 853 in Adolescents With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20090223
Record Dates: First submitted 2010-04-22; First posted 2010-06-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
Keywords: Amgen; Adolescent; Safety
MeSH Terms: conditions — Asthma | interventions — vidupiprant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- AMG 853 (Experimental)
  Interventions: Drug: AMG 853
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 853 — Single dose administration of AMG 853 or placebo in tablet form to adolescent and adult subjects with asthma
  Arms: AMG 853
Drug: Placebo — Placebo to AMG 853
  Arms: Placebo

SUMMARY:
The purpose of this study is to study the safety and tolerability in adolescent and adult subjects with intermittent or mild to moderate persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects ≥12 to < 18 years of age (for Cohorts 1, 2, and 3 as indicated in the study design).
* Male and/or non-reproductive female subjects between 18 and 50 years of age, inclusive (for cohort 4).
* Females of non-reproductive potential must have documented medical history (ie, postmenopausal by history - no menses for 1 year - and follicle-stimulating hormone value (FSH) consistent with postmenopausal status per laboratory ranges; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy).
* Females of child-bearing potential and females who cannot document non-reproductive potential must agree to use highly effective methods of birth control for the duration of the study and for 2 weeks after study drug administration. Males whose partners are of child bearing potential must agree to use highly effective methods of birth control for the duration of the study and continuing for 12 weeks after study drug administration. Highly effective methods of birth control (i.e., those with a failure rate of less than 1% per year) include sexual abstinence (males, females), vasectomy or a condom supplemented with the use of a spermicide (males) and occlusive cap (diaphragm or cervical/vault caps), hormonal birth control, or intrauterine device (IUD) used by the female partner.
* Male subjects whose partners become pregnant during the study must practice sexual abstinence or use a condom with spermicide for two weeks following study drug administration to ensure the unborn child is not potentially exposed to AMG 853 via semen. The pregnant partner information will be reported to Amgen per the Pregnancy Notification Worksheet.
* Intermittent or mild to moderate persistent asthma for the past 3 months (as defined by the 2004 Global Initiative for Asthma [GINA] guidelines).
* On a stable pharmacologic regimen for the treatment of asthma for at least 3 months prior to study enrollment and does not anticipate any change to the regimen during the course of the study.
* Forced Expiry Volume in 1 second (FEV1) at screening visit ≥ 70% of predicted normal value (without aid of bronchodilator).
* FEV1 reversibility greater than or equal to 12% from baseline within 30 minutes of inhaled (up to 400 μg) or nebulized (up to 5 mg) albuterol at the office screening visit. Subjects unable to demonstrate reversibility during screening, must provide the most recent evidence of documented reversibility to the Amgen Medical Monitor and the principal investigator for review.
* Clinically acceptable physical examination, electrocardiogram (ECG), and clinical laboratory test values for the population tested. Any abnormal clinical laboratory results and/or ECG values must be discussed with the Sponsor.

Exclusion Criteria:

* History or evidence of clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Experienced an asthma exacerbation (defined as a disease episode resulting in treatment in an emergency room or urgent care facility, or an episode treated with oral corticosteroids) during the 3 months prior to study enrollment.
* Hospitalized for asthma during the 6 months prior to study enrollment; or ever intubated for the treatment of asthma.
* Use of oral corticosteroids within 3 months prior to study enrollment.
* Evidence of recent (within 2 weeks of study enrollment) or current signs or symptoms of an upper respiratory infection (eg, viral, bacterial).
* Known positive tuberculin skin test (if not treated with appropriate chemoprophylaxis) or untreated exposure to a patient with active tuberculosis.
* History of autoimmune disorder (eg, rheumatoid arthritis, systemic lupus).
* Creatinine clearance within the screening period of less than 80 mL/min as calculated by the Cockcroft-Gault method.
* History of clinically significant cardiovascular, renal, hepatic or respiratory disease other than asthma.
* History suggestive of esophageal, gastric, or duodenal ulceration or bowel disease (including but not limited to peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease or irritable bowel syndrome), or a history of gastrointestinal surgery (excluding uncomplicated appendectomy).
* Any positive test for cotinine (tobacco use) on the day before dosing. A positive cotinine level is defined as any level exceeding the upper limit of normal as per local laboratory reference ranges.
* Known substance abuse (eg, alcohol, licit or illicit drugs) within 1 year of dosing as defined by Diagnostic and Statistical Manual version 4, text revsion (DSM-IV-TR) criteria.
* Any positive test for drugs and or alcohol use on the day before dosing (day -1). For subjects of legal drinking age, alcohol should not be consumed within 48 hours of day -1 and throughout the study. Alcohol use is not permitted for subjects below the legal drinking age.
* Positive pregnancy test at screening or day -1.
* Females who are lactating or breastfeeding.
* with pregnant partners.
* Inability or unwillingness to swallow tablets.
* A history of malignancy of any type, other than surgically excised non-melanomatous skin cancers or in situ cervical cancer within 5 years before the day of dosing.
* Donated greater than 500 mL of blood or blood products within 60 days of dosing.
* Subjects who have received any investigational drug (or have used an investigational device) within the 30 days before receiving the first dose of study medication, or at least 5 elimination half-lives (whichever is longer).
* Subjects who were previously exposed to AMG 853.
* Use of any prescription (eg, angiotensin inhibitors) or non-prescription [eg, non-steroidal anti-inflammatory drugs (NSAIDS)] medications including asthma medications (eg, inhaled cromolyn, inhaled ipratropium, inhaled tiotropium, theophylline) within 7 days of study start with the exception of inhaled corticosteroid therapy (≤ 660 μg/day fluticasone or ≤ 480 μg/day beclomethasone, or equivalent), inhaled short-acting and long-acting β-2 agonists, and montelukast.
* Use of any over-the-counter or prescription medications (specifically including, but not limited to antacids, H2- blockers, and proton pump inhibitors, aspirin or other NSAIDS within 28 days of dosing. Acetaminophen (up to 2 g per day) for analgesia and hormone replacement therapy (eg, estrogen) will be allowed.
* Use of any known inhibitors of CYP3A4/P-gp such as ketoconazole, itraconazole, HIV protease inhibitors, nefazadone, cyclosporine, erythromycin, clindamycin, tetracycline, and clarithromycin within 14 days or 5 half lives, whichever is longer; or grapefruit juice or grapefruit containing products within 7 days prior to investigational product administration.
* Use of any known CYP inducers such as rifampin, oral corticosteroids, or anticonvulsants within 30 days or 5 half-lives, whichever is longer, before investigational product administration.
* All herbal medicines (eg, St. John's Wort), vitamins, and supplements consumed by the subject within 30 days prior to the first dose of investigational product, and continued use if appropriate, will be reviewed by the Principal Investigator and the Amgen Medical Monitor.
* History of hypersensitivity or allergic reaction to sulfonamide drugs.
* Positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen, or hepatitis C antibodies.
* Known history of Gilbert's syndrome.
* Unwilling or unable to return to the research facility for follow-up assessments as required per protocol.
* Any other condition that might reduce the chance of obtaining data (eg, known poor compliance) required by the protocol or that might compromise the ability to give truly informed consent.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of treatment-emergent adverse events, safety and laboratory assessments in adolescent subjects with intermittent or mild to moderate asthma as a measure of safety and tolerability | Throughout the study duration

SECONDARY OUTCOMES:
Pharmacokinetic parameters (including Cmax and AUC) for a single dose administration of AMG 853 in adolescent and adult subjects | Throughout study duration (at predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 168 hours after dose)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com